CLINICAL TRIAL: NCT00452517
Title: Comparison of Stent Graft, Sirolimus Stent, and Bare Metal Stent Implanted in Patients With Acute Coronary Syndrome: Clinical and Angiographic Follow-up
Brief Title: Comparison of Stent Graft, Sirolimus Stent, and Bare Metal Stent Implanted in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SG-SIR-BM-07
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2007-03-27 (Estimated); Status verified 2007-03

CONDITIONS: Acute Coronary Syndrome
Keywords: bare metal stents; sirolimus-eluting stents; coronary polytetrafluoroethylene stent graft; acute coronary syndrome; quantitative coronary angiography analysis; major adverse cardiac events; in-stent restenosis; target lesion revascularisation
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention

SUMMARY:
During the 6-month period 119 patients with acute coronary syndrome, were randomized to either stent graft group (n=40), sirolimus eluting stent group (n=39), or bare metal stent group (n=40). Demographic, angiographic and procedural characteristics were similar for all three groups. The incidence of 6-month major adverse coronary events were analysed.

DETAILED DESCRIPTION:
Background: Percutaneous coronary intervention with stent implantation is a standard therapy for patients with acute coronary syndrome. The in-stent restenosis is still a problem. Recently, drug eluting stents reduce the incidence of this unfavorable event. The primary role of the polytetrafluoroethylene stent graft (PTFE) is management of coronary perforations, closure of coronary aneurysms, and in degenerated saphenous vein grafts. We compared these stents in native coronary vessels in patients with acute coronary syndrome with sirolimus and bare metal stents, for possible reduction of in-stent restenosis.

Methods and results: During the 6-month period 119 patients with acute coronary syndrome, were randomized to either stent graft group (n=40), sirolimus eluting stent group (n=39), or bare metal stent group (n=40). Demographic, angiographic and procedural characteristics were similar for all three groups. The incidence of 6-month major adverse coronary events was similar in all three groups. The target lesion revascularisation was higher in the bare metal stent group (P=0.044). The primary end-point, restenosis rate at six-month follow-up was higher in the bare metal stent group, compared with the stent graft and sirolimus eluting stent groups. The percent diameter stenosis in follow-up was significantly higher in bare metal stent group (P=0.005). The late loss was significantly lower in the sirolimus eluting stent group (0.23 mm), compared with the bare metal stent group (P= 0.034). There was a trend of lower late loss in the stent graft group, compared with bare metal stent group.

Conclusion: Three groups of stents implanted in patients with acute coronary syndrome (stent-graft, sirolimus and bare metal), did not differ regarding the incidence of major adverse cardiac events. Sirolimus-eluting stents had a lower incidence of in-stent restenosis in comparison with bare metal stent group. Stent graft implanted in native coronary arteries appears to be safe and efficient in patients with acute coronary syndrome, but a significant reduction of in-stent restenosis was not achieved.

ELIGIBILITY:
Inclusion Criteria:

* stent implantation in acute coronary syndrome

Exclusion Criteria:

* previous percutaneous coronary intervention or coronary artery bypass graft surgery
* multivessel, diffuse disease, tortuous vessel
* arteries less than 3 mm in diameter
* distal stenosis location
* left main and bifurcation lesions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-03; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Three groups of stents implanted in patients with acute coronary syndrome (stent-graft, sirolimus and bare metal), did not differ regarding the incidence of major adverse cardiac events.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Strozzi, MD, Principal Investigator — University hospital Zagreb
Locations (1):
- University hospital Zagreb, Zagreb, Croatia

REFERENCES:
- [Background] Keeley EC, Boura JA, Grines CL. Comparison of primary and facilitated percutaneous coronary interventions for ST-elevation myocardial infarction: quantitative review of randomised trials. Lancet. 2006 Feb 18;367(9510):579-88. doi: 10.1016/S0140-6736(06)68148-8. PMID 16488801
- [Background] Saia F, Lemos PA, Lee CH, Arampatzis CA, Hoye A, Degertekin M, Tanabe K, Sianos G, Smits PC, McFadden E, Hofma SH, van der Giessen WJ, de Feyter PJ, van Domburg RT, Serruys PW. Sirolimus-eluting stent implantation in ST-elevation acute myocardial infarction: a clinical and angiographic study. Circulation. 2003 Oct 21;108(16):1927-9. doi: 10.1161/01.CIR.0000096053.87580.CD. Epub 2003 Oct 13. PMID 14557354
- [Derived] Strozzi M, Anic D. Comparison of stent graft, sirolimus stent, and bare metal stent implanted in patients with acute coronary syndrome: clinical and angiographic follow-up. Croat Med J. 2007 Jun;48(3):348-52. PMID 17589978